CLINICAL TRIAL: NCT02443883
Title: Randomized Phase 2 Trial Evaluating Pharmacokinetics and Safety of Four Ramucirumab Dosing Regimens in Second-Line Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Phase 2 Study of Ramucirumab (LY3009806) in Participants With Gastric or Gastroesophageal Junction (GEJ) Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15608; I4T-MC-JVDB (Other: Eli Lilly and Company); 2014-003791-23 (EudraCT Number)
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2019-07

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ramucirumab Regimen 1 (Experimental): Standard dose of 8 milligram per kilogram (mg/kg) ramucirumab given intravenously (IV) on day 1 and day 15 of each cycle (28-day cycle) until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab
- Ramucirumab Regimen 2 (Experimental): Experimental dose of 12 mg/kg ramucirumab given IV on day 1 and day 15 of each cycle (28-day cycle) until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab
- Ramucirumab Regimen 3 (Experimental): Experimental dose of 6 mg/kg ramucirumab given IV on day 1, 8, 15 and 22 of each cycle (28-day cycle) until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab
- Ramucirumab Regimen 4 (Experimental): Experimental dose of 8 mg/kg ramucirumab given IV on day 1 and day 8 of each cycle (21-day cycle) until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B

SUMMARY:
The main purpose of this study was to evaluate the safety and pharmacokinetics of administering various dose regimens of ramucirumab in participants with advanced gastric cancer whose disease has progressed during or following prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a histopathologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction (GEJ).
* The participant has documented disease progression during or within 4 months after the last dose of first-line chemotherapy for metastatic disease, or during or within 6 months after the last dose of neoadjuvant or adjuvant therapy.
* The participant received combination chemotherapy prior to disease progression.

  * Prior chemotherapy regimens must include a platinum and/or a fluoropyrimidine component and must not include a taxane or antiangiogenic agent.
* The participant has metastatic disease or locally advanced disease that is measurable or nonmeasurable, but is evaluable disease by radiological imaging per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
* Patients are eligible if they are considered not appropriate, for whatever reason, for treatment with ramucirumab in combination with paclitaxel.
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The participant has adequate organ function, including:

  * Total bilirubin 1.5 × the upper limit of institutional normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 3 × ULN. If the liver has tumor involvement, AST and ALT <5 × ULN are acceptable.
  * Serum creatinine 1.5 × ULN or calculated creatinine clearance (per the Cockcroft-Gault formula or equivalent and/or 24-hour urine collection) 60 milliliters/minute (mL/min).
  * Urinary protein is <2+ on dipstick or routine urinalysis.
  * Absolute neutrophil count 1.5 × 10^9/Liter (L), platelets 100 × 10^9/L, and hemoglobin 9 g/deciliter (dL) (5.58 millimoles/Liter).
  * International normalized ratio 1.5 × ULN or prothrombin time 5 seconds above ULN.
  * Partial thromboplastin time 5 seconds above ULN.
* The participant has an estimated life expectancy of 12 weeks in the judgment of the investigator.
* The participant, if female and of child-bearing potential, must have a negative serum or urine pregnancy test within 7 days prior to randomization.

Exclusion Criteria:

* The participant has squamous cell or undifferentiated gastric cancer.
* The participant is receiving chronic therapy with any of the following within 7 days prior to randomization:

  * Nonsteroidal anti-inflammatory agents (NSAIDs; such as indomethacin, ibuprofen, naproxen, or similar agents), or
  * Other anti-platelet agents (such as clopidogrel, ticlopidine, dipyridamole, or anagrelide). Aspirin use at doses up to 325 milligrams (mg)/day is permitted.
* The participant received radiotherapy within 14 days prior to randomization.
* The participant received >1 line of prior therapy for the treatment of locally advanced and unresectable or metastatic gastric or GEJ (Siewert Types I-III) adenocarcinoma.
* The participant received previous treatment with agents targeting the vascular endothelial growth factor (VEGF)/VEGF receptor 2 signaling pathway.
* The participant has documented brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression.
* The participant experienced any arterial thromboembolic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization.
* The participant has symptomatic congestive heart failure (New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
* The participant has uncontrolled hypertension, as defined in Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, prior to initiating study treatment, despite antihypertensive intervention.
* The participant underwent major surgery within 28 days prior to randomization or central venous access device placement within 7 days prior to randomization.
* The participant has a history of gastrointestinal perforation or fistula within 6 months prior to randomization.
* The participant has any condition (for example, psychological, geographical, or medical) that does not permit compliance with the study and follow-up procedures or suggests that the participant is, in the investigator's opinion, not an appropriate candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (5):
  - Arizona Clinical Research Center, Tucson, Arizona
  - USC Norris Cancer Hospital, Los Angeles, California
  - Carolinas Medical Center, Charlotte, North Carolina
  - Oklahoma Cancer Specialists & Research Institute, LLC, Tulsa, Oklahoma
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viedma
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingswood
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- New Zealand (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auckland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
- Russia (4):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - Leningrad regional clinical hospital, Saint Petersburg
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Košice
- Turkey (Türkiye) (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fatih
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medreseboğazı
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pendik
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cardiff
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Exeter
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completion was defined as death due to any cause or disease progression.
Groups:
- Ramucirumab Regimen 1: Ramucirumab (8milligram per kilogram [mg/kg]) given intravenously (IV) on day 1 and day 15 of each cycle (28-day cycle) until discontinuation criteria are met.
- Ramucirumab Regimen 2: Ramucirumab (12 mg/kg) given IV on day 1 and day 15 of each cycle (28-day cycle) until discontinuation criteria are met.
- Ramucirumab Regimen 3: Ramucirumab (6 mg/kg) given IV on day 1, 8, 15 and 22 of each cycle (28-day cycle) until discontinuation criteria are met.
- Ramucirumab Regimen 4: Ramucirumab (8 mg/kg) given IV on day 1 and day 8 of each cycle (21-day cycle) until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Ramucirumab Regimen 1 | Ramucirumab Regimen 2 | Ramucirumab Regimen 3 | Ramucirumab Regimen 4
Started | 40 | 42 | 41 | 41
Received at Least One Dose of Study Drug | 38 | 42 | 41 | 40
Completed | 34 | 38 | 40 | 36
Not Completed | 6 | 4 | 1 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2
Not completed — Randomized, but never treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ramucirumab Regimen 1: Ramucirumab (8 mg/kg) given IV on day 1 and day 15 of each cycle (28-day cycle) until discontinuation criteria are met.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab Regimen 1 | Ramucirumab Regimen 2 | Ramucirumab Regimen 3 | Ramucirumab Regimen 4 | Total
Number analyzed (Participants) | 40 | 42 | 41 | 41 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (14.0) | 58.7 (10.4) | 60.5 (12.3) | 56.2 (12.9) | 58.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 6 | 9 | 36
  Male | 29 | 32 | 35 | 32 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 6 | 7 | 22
  Not Hispanic or Latino | 32 | 37 | 33 | 32 | 134
  Unknown or Not Reported | 2 | 2 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 32 | 35 | 35 | 33 | 135
  More than one race | 6 | 7 | 5 | 6 | 24
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 2 | 1 | 1 | 3 | 7
  Argentina | 5 | 1 | 2 | 6 | 14
  Romania | 4 | 6 | 10 | 7 | 27
  Turkey | 3 | 4 | 2 | 2 | 11
  Hungary | 0 | 3 | 3 | 1 | 7
  United States | 2 | 3 | 2 | 1 | 8
  Poland | 6 | 6 | 7 | 5 | 24
  United Kingdom | 7 | 10 | 8 | 6 | 31
  Slovakia | 3 | 1 | 2 | 1 | 7
  Australia | 1 | 2 | 0 | 5 | 8
  France | 1 | 1 | 2 | 1 | 5
  Russia | 6 | 4 | 2 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Description: The Cmin is the minimum observed serum concentration of ramucirumab.
Time Frame: Day 29, 43, 71 and 85: predose
Population: All randomized participants who received at least one dose of ramucirumab and had evaluable ramucirumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Ramucirumab Regimen 1 | Ramucirumab Regimen 2 | Ramucirumab Regimen 3 | Ramucirumab Regimen 4
Number analyzed (Participants) | 38 | 42 | 41 | 40
microgram per milliliter (µg/mL)
  Day 29: number analyzed (Participants) | 29 | 32 | 28 | 31
  Day 29 | 32.9 (51) | 59.5 (60) | 69.3 (45) | 71.6 (37)
  Day 43: number analyzed (Participants) | 15 | 22 | 18 | 17
  Day 43 | 47.6 (36) | 71.0 (58) | 83.0 (57) | 57.4 (44)
  Day 71: number analyzed (Participants) | 6 | 12 | 12 | 10
  Day 71 | 60.4 (34) | 65.0 (60) | 122 (65) | 97.1 (46)
  Day 85: number analyzed (Participants) | 6 | 10 | 11 | 9
  Day 85 | 64.3 (40) | 79.4 (46) | 125 (56) | 81.6 (50)

2. Secondary Outcome: Immunogenicity: Number of Participants With Anti-Ramucirumab Antibodies
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies was summarized by treatment group. A treatment-emergent anti-drug antibodies (TEADA) sample was defined as: a post treatment sample with at least a 4-fold increase in titer from pre treatment sample; or 1:20 post treatment titer for participants that had no detectable ADA titer at baseline.
Time Frame: Predose Cycle 1 Through Short Term Follow Up (Up to 5 Months)
Population: All randomized participants who received at least 1 dose of ramucirumab and had evaluable anti-ramucirumab antibody measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab Regimen 1 | Ramucirumab Regimen 2 | Ramucirumab Regimen 3 | Ramucirumab Regimen 4
Number analyzed (Participants) | 19 | 26 | 20 | 22
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Rate of Progression Free Survival (PFS) at the First 6-Week Tumor Assessment
Description: PFS defined as the time from first day of therapy to first evidence of disease progression per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) or death from any cause up to the first 6-week tumor assessment. Progressive Disease (PD) is at least 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study and absolute increase of at least 5 mm.Appearance of 1 or more new lesions was also considered progression. Nontarget PD is unequivocal progression of existing nontarget lesions.Appearance of 1 or more new nontarget lesions was also considered PD.Participants with no baseline disease assessment: PFS time was censored at the randomization date,regardless of whether or not objectively determined disease progression or death has been observed.
Time Frame: Baseline until the first 6-week tumor assessment
Population: All randomized participants.Censored participants:Ramucirumab Regimen 1 = 8,Ramucirumab Regimen 2 =10,Ramucirumab Regimen 3=8 and Ramucirumab Regimen 4=12. PFS survival rate at the first 6-week assessment was estimated using the Kaplan-Meier method which takes into consideration who were censored prior to 6 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ramucirumab Regimen 1 | Ramucirumab Regimen 2 | Ramucirumab Regimen 3 | Ramucirumab Regimen 4
Number analyzed (Participants) | 40 | 42 | 41 | 41
Percentage of participants | 43.9 [27.3 to 59.3] | 61.9 [44.9 to 75.0] | 53.0 [36.2 to 67.3] | 51.2 [34.2 to 65.9]

ADVERSE EVENTS:
Time Frame: Up To 3 Years and 3 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Ramucirumab Regimen 1 | Ramucirumab Regimen 2 | Ramucirumab Regimen 3 | Ramucirumab Regimen 4
Serious Adverse Events (participants affected / at risk) | 10/38 | 11/42 | 10/41 | 18/40
Other Adverse Events (participants affected / at risk) | 30/38 | 31/42 | 36/41 | 31/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab Regimen 1 (N=38) | Ramucirumab Regimen 2 (N=42) | Ramucirumab Regimen 3 (N=41) | Ramucirumab Regimen 4 (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 4 (5)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thoracic cavity drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab Regimen 1 (N=38) | Ramucirumab Regimen 2 (N=42) | Ramucirumab Regimen 3 (N=41) | Ramucirumab Regimen 4 (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 (12) | 5 (15) | 5 (11) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 10 (14) | 7 (9) | 4 (8)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (8) | 7 (7) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 9 (12) | 4 (5) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (9) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4) | 4 (5) | 7 (9)
Vomiting (Gastrointestinal disorders) | 6 (8) | 6 (7) | 8 (13) | 7 (10)
Asthenia (General disorders) | 2 (2) | 3 (3) | 4 (8) | 3 (4)
Early satiety (General disorders) | 0 (0) | 3 (6) | 0 (0) | 1 (1)
Fatigue (General disorders) | 10 (12) | 12 (17) | 6 (7) | 9 (9)
Oedema peripheral (General disorders) | 1 (1) | 4 (5) | 2 (2) | 2 (3)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 4 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 5 (7) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 5 (8) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 5 (5) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (4) | 2 (2) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 9 (16) | 11 (13) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (4) | 1 (2) | 4 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 3 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (3) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (5) | 1 (2) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (8) | 6 (8) | 5 (8) | 3 (3)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (5) | 1 (1) | 2 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (6) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 6 (7) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 6 (8) | 2 (3) | 7 (8) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less